CLINICAL TRIAL: NCT00766519
Title: Effect of Intraoperative Volume Optimization on Outcome After Intrabdominal Surgery: a Multicenter, Randomized, Double-blind, Comparative Study
Brief Title: Effect of Intraoperative Volume Optimization on Outcome After Intrabdominal Surgery
Acronym: EVOLUTION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007-A01436-47; PHRC 2006/1915 (Other: DHOS); 2007/0723 (Other: sponsor)
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Hemodynamic Instability; Surgery
Keywords: fluid responsiveness; monitoring; arterial pulse pressure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Optimization (Experimental): volume optimization: continuous monitoring of the respiratory-induced arterial pulse pressure variation during surgery and systematic minimization to 10% or less by volume loading
  Interventions: Other: volume optimization
- control; standard volume administration (Active Comparator): standard volume administration
  Interventions: Other: standard volume administration

INTERVENTIONS:
Other: volume optimization — Fluid management:
  * basal fluid administration = 5 ml/kg/h lactated Ringer's solution
    + systematic minimization of the arterial pulse pressure variation (PPV) to 10% or less by volume loading (6% hydroxyethyl starch) throughout surgery
  * hypovolemia suspected : fluids (1. crystalloids, 2. 6% hydroxyethyl starch) only if PPV is > 10%
  Other Names: preload optimization
  Arms: Optimization
Other: standard volume administration — Fluid management:
  * basal fluid administration = 5 ml/kg/h lactated Ringer's solution
  * hypovolemia suspected : fluids (1. crystalloids, 2. 6% hydroxyethyl starch) according to predetermined algorithm primarily based on mean arterial pressure, heart rate, and urine output, and secondary on PPV
  Other Names: fluid compensation
  Arms: control; standard volume administration

SUMMARY:
The purpose of this study is to determine whether intraoperative goal-directed fluid management (with goal = cardiac stroke volume maximization) based on respiratory-induced pulse pressure variation monitoring may improve outcome after intrabdominal surgery

DETAILED DESCRIPTION:
Recent studies strongly suggest that intraoperative oesophageal doppler guided fluid management may improve outcome after intrabdominal surgery. In these studies, however, the number of patients was often small, and management in control groups as well as postoperative complications were usually not precisely defined. In addition, widespread use of oesophageal doppler cannot be advocated in routine surgery, and the strategy necessitates repeated volume loading. This may lead to unnecessary intravenous fluids which may be deleterious, and intraoperative fluid restriction has also been shown to improve clinical outcome. In this context, indices reflecting the hemodynamic changes during mechanical ventilation (the so-called "dynamic indices", and more specifically the respiratory-induced pulse pressure variation) have been shown to accurately predict fluid responsiveness in mechanically ventilated patients. Automated and continuous calculation of pulse pressure variation variation from standard peripheral (typically radial) arterial line has recently been validated. This study was thus designed to determine whether intraoperative goal-directed fluid management (with goal = cardiac stroke volume maximization) based on pulse pressure variation monitoring would improve outcome after intrabdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* major elective intrabdominal surgery

Exclusion Criteria:

* arrhythmia
* hepatectomy
* associated thoracic surgery
* laparoscopy
* pregnancy
* allergy to colloid solution or anesthesia protocol
* arterial catheter not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Total number of patients with complications | first 7 postoperative days

SECONDARY OUTCOMES:
total number of complications | first 7 postoperative days
SOFA (Sequential Organ Failure Assessment) score | postoperative days 1 and 5
Time to initial passage of flatus and feces | postoperative
duration of stay in intensive care unit | postoperative
Duration of hospital stay | postoperative
death | in-hospital and postoperative day 28
volumes of fluid administered | duration of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Benoit TAVERNIER, MD, PhD, Study Director — University Hospital, Lille; Benoit VALLET, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (6):
- France (6):
  - University Hospital, Amiens
  - University Hospital, Caen
  - Département d'Anesthésie-Réanimation, Hôpital Estaing, CHU, Clermont-Ferrand
  - University hospital Henri-Mondor, Créteil
  - University Hospital, Lille
  - University Hospital, Rouen